CLINICAL TRIAL: NCT01144923
Title: Randomized, Comparative-effectiveness Study Comparing Epidural Steroid Injections to Conservative Management With Medications and Physical Therapy in Patients With Cervical Radiculopathy
Brief Title: Conservative Therapy Versus Epidural Steroids for Cervical Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Steven P. Cohen, Professor, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00036062
Record Dates: First submitted 2010-06-14; First posted 2010-06-16 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Cervical Radiculopathy
Keywords: epidural steroid injection; neck pain; pharmacotherapy; radiculopathy
MeSH Terms: conditions — Radiculopathy; Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Conservative treatment (Active Comparator): Pharmacotherapy with nortriptyline and/ or gabapentin, physical therapy (e.g. range of motion, therapeutic massage, strengthening exercises), and possibly others (e.g. acupuncture)
  Interventions: Other: Gabapentin and/or Nortriptyline, Physical therapy
- Epidural Steroids (Experimental): A series of up to 3 epidural steroid injections (ESI)with depo-methylprednisolone
  Interventions: Procedure: Epidural Steroid Injections (ESI)
- Combination Treatment (Experimental): These patients will receive both treatments. They can have up to 3 epidural steroid injections (ESI) with depo-methylprednisolone, and conservative treatment (i.e. pharmacotherapy with nortriptyline and/ or gabapentin, and physical therapy)
  Interventions: Other: Combination treatment

INTERVENTIONS:
Other: Gabapentin and/or Nortriptyline, Physical therapy — Nortriptyline up to 125 mg po qhs, and / or Gabapentin up to 1200 mg po q8h, Physical therapy (e.g. range of motion, strengthening, therapeutic massage, TENS)
  Arms: Conservative treatment
Procedure: Epidural Steroid Injections (ESI) — Series of up to 3 cervical epidural steroid injections (ESI) with depo-methylprednisolone
  Arms: Epidural Steroids
Other: Combination treatment — Series of up to 3 cervical epidural steroid injections with depo- methylprednisolone plus Nortriptyline up to 125 mg po qhs and /or Gabapentin up to 1200 mg po q8h, and Physical therapy (e.g. TENS, exercise, range of motion)
  Arms: Combination Treatment

SUMMARY:
The main objective of this study is to determine whether interventional treatment (i.e. epidural steroids), conservative therapy, or the combination, is superior for cervical radiculopathy. One hundred and sixty eight patients with radicular neck pain will be randomized in a 1:1:1 ratio to receive either cervical epidural steroid injections (CESI), non-interventional management with physical therapy and medications, or a combination of the two. The first follow-up visit will be at 1-month. In patients who obtain some benefit but continue to report significant pain, either a 2nd CESI can be done, the patient's medications can be adjusted, or both in the combination group. Those patients who fail to obtain any benefit will exit the study to receive another treatment or alternative care. The second follow-up visit will be at 3-months. Similar to the 1-month follow-up, the doctor may elect to change nothing in patients who are satisfied, adjust medications, schedule the patient for another CESI, or do both in the combination group. Patients who fail to obtain any benefit can exit the study to receive alternative treatment. The final follow-up visit will be at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Cervical radicular pain based on history and physical exam (e.g. pain radiating into one or both extremities, sensory loss, muscle weakness, Spurling's test etc.)
2. NRS arm pain score > 3
3. MRI evidence of disc pathology consistent with symptoms

Exclusion Criteria:

1. Untreated coagulopathy
2. Previous spine surgery
3. No MRI study
4. Arm pain > 4 years duration
5. Epidural steroid injection within past 3 years
6. Radiculopathy not resulting from disc pathology (e.g. foraminal stenosis or tumor)
7. Signs or symptoms or myelopathy or spinal cord compression
8. Previous failed trials with gabapentin or pregabalin, and nortriptyline or amitriptyline
9. Allergic reactions to gabapentin or nortriptyline
10. Referrals from surgery for diagnostic injections for surgical evaluation
11. Serious medical (e.g. congestive heart failure) or psychiatric (untreated depression) condition that might preclude optimal outcome
12. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
numerical rating scale (NRS) arm pain scores | 1 month after treatment
  arm pain on a 0-10 scale

SECONDARY OUTCOMES:
NRS Arm pain | 3 months
  0-10 scale
NRS arm pain | 6 months
  0-10 scale
NRS neck pain | 1- month
  0-10 scale
NRS neck pain | 3 months
  0-10 scale
NRS neck pain | 6 months
  0-10 scale
medication reduction | 1-6 months
  Cessation of non-opioid analgesic and/ or > 20% decrease in opioid consumption
Global perceived effect | 1-6 months
  categorical variable assessing "satisfaction" with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Study Director — Johns Hopkins University; Salim Hayek, MD, PhD, Principal Investigator — Case Western; Rick Fisher, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins Medical Institutions, Baltimore, Maryland

REFERENCES:
- [Background] Hogg-Johnson S, van der Velde G, Carroll LJ, Holm LW, Cassidy JD, Guzman J, Cote P, Haldeman S, Ammendolia C, Carragee E, Hurwitz E, Nordin M, Peloso P; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. The burden and determinants of neck pain in the general population: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S39-51. doi: 10.1097/BRS.0b013e31816454c8. PMID 18204398
- [Background] Carragee EJ, Hurwitz EL, Cheng I, Carroll LJ, Nordin M, Guzman J, Peloso P, Holm LW, Cote P, Hogg-Johnson S, van der Velde G, Cassidy JD, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Treatment of neck pain: injections and surgical interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S153-69. doi: 10.1097/BRS.0b013e31816445ea. PMID 18204388
- [Background] Hurwitz EL, Carragee EJ, van der Velde G, Carroll LJ, Nordin M, Guzman J, Peloso PM, Holm LW, Cote P, Hogg-Johnson S, Cassidy JD, Haldeman S; Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Treatment of neck pain: noninvasive interventions: results of the Bone and Joint Decade 2000-2010 Task Force on Neck Pain and Its Associated Disorders. Spine (Phila Pa 1976). 2008 Feb 15;33(4 Suppl):S123-52. doi: 10.1097/BRS.0b013e3181644b1d. PMID 18204386